CLINICAL TRIAL: NCT01529918
Title: e-Diabetes:Uptake, Patient Preferences and Clinical Outcomes Regarding Self-screening and Clinical Follow-up Using Web-based Technologies in a Large Team-based Primary Care Setting
Brief Title: Detecting Diabetes Sooner With a Risk Survey for the Family Doctor:Comparing Internet and Traditional Methods of Communication for Patients and Doctors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: eDM-1
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2009-10

CONDITIONS: Diabetes
Keywords: Diabetes; Self-screening; Web-based technology; follow-up clinical care; randomized control trial
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- web-intervention group (Experimental): Participants will receive access to the CAN-RISK (Canadian Diabetes Risk Assessment) questionnaire either via personal patient electronic health record or an online version
  Interventions: Other: CANRISK (Canadian Diabetes Association Assessment)
- paper-based group (No Intervention): Participants allocated to paper-based will receive the CAN-RISK questionnaire for diabetes risk-assessment via paper-based
  Interventions: Other: CANRISK (Canadian Diabetes Association Assessment)

INTERVENTIONS:
Other: CANRISK (Canadian Diabetes Association Assessment) — Self-risk assessment questionnaire for diabetes

SUMMARY:
This pilot RCT study aims to develop and evaluate the uptake, feasibility, and potential value of a strategy for web-diabetes risk assessment versus paper-based methods in an undiagnosed diabetes population over 40 years of age from all listed FHT provided through an electronic medical record database. Following randomization, intervention participants will have the option to decide to use web-based self-screening and the control group will receive only a paper-based method. There will be two options for web-based screening; one involves completion of the CAN-RISK screening tool as part of a personal health record self-management program (MyOscar) versus a one off online risk-assessment. The intervention and control group will be compared with respect to risk-assessment uptake. Educational sessions and further assessment of diabetes conducted by the clinical health care team will be offered to all participants who scored a high risk of diabetes in accordance with the CAN-RISK results. Actual numbers of diabetes cases in those with a high risk score will be compared between the intervention and control groups as well as compared to the usual method of diabetes screening in a randomly chosen non-identifiable sample from the same clinical setting in the same one year period. The assessment of patient acceptability in feasibility of the implementation of the self-screening tool will be accomplished through surveys designed to be completed by patients and staff.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 and over who did not have diagnosis of diabetes and no previous use of personal health record (MyOscar)

Exclusion Criteria:

* People with diabetes, and those who are already registered as MyOSCAR (personal e-health record) users

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Patient's uptake and preferences | 1 year
  Numbers of patients participating in the self risk-assessment, and a comparison of paper versus web-based technologies will be collected.
  * Demographics of the 2 groups will be compared.
  * A user-satisfaction survey will assess patients' perceptions of the technologies. Use of necessary qualitative techniques can be considered as well.

SECONDARY OUTCOMES:
The comparison of yield of actual diabetes detected from those who have high risk at self risk-assessment, compared to the usual diabetes detection rate in a random sample from the practice within a one year period. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gina Agarwal, Dr., Principal Investigator — McMaster University, Department of Family Medicine